CLINICAL TRIAL: NCT04338269
Title: A Phase III, Multicenter, Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Atezolizumab Given in Combination With Cabozantinib Versus Cabozantinib Alone in Patients With Inoperable, Locally Advanced, or Metastatic Renal Cell Carcinoma Who Experienced Radiographic Tumor Progression During or After Immune Checkpoint Inhibitor Treatment
Brief Title: A Study of Atezolizumab in Combination With Cabozantinib Compared to Cabozantinib Alone in Participants With Advanced Renal Cell Carcinoma After Immune Checkpoint Inhibitor Treatment
Acronym: CONTACT-03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Exelixis (Industry); Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO41994
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — atezolizumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezo+Cabo (Experimental): Participants will receive atezolizumab every 3 weeks on Day 1 of each 21-day cycle (1 cycle=21 days) plus oral tablets of cabozantinib every day.
  Interventions: Drug: Atezolizumab; Drug: Cabozantinib
- Cabozantinib (Active Comparator): Participants will receive cabozantinib every day.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be administered at a fixed dose on Day 1 of each 21-day cycle by IV infusion every 3 weeks.
  Other Names: Tecentriq
  Arms: Atezo+Cabo
Drug: Cabozantinib — Cabozantinib 60 mg (three 20-mg tablets) administered orally once daily.
  Other Names: Cabometyx

SUMMARY:
This is a Phase III, multicenter, randomized, open-label study designed to evaluate the efficacy and safety of atezolizumab given in combination with cabozantinib versus cabozantinib alone in participants with inoperable, locally advanced, or metastatic renal cell carcinoma (RCC) who experienced radiographic tumor progression during or after Immune Checkpoint Inhibitor (ICI) treatment in the metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic clear cell or non-clear cell (papillary, chromophobe, and unclassified only) RCC. RCC with sarcomatoid features is allowed. Patients with the chromophobe subtype of non-clear cell RCC must have sarcomatoid differentiation.
* Radiographic disease progression to prior ICI therapy for RCC. Patients who experienced radiographic tumor progression during or within 6 months after the last dose of adjuvant ICI are also eligible. ICI is defined by anti-PD-L1 or anti-PD1 antibody including atezolizumab, avelumab, pembrolizumab, durvalumab, or nivolumab. Only patients for whom the immediate preceding line of therapy was an ICI are allowed.
* Measurable disease per RECIST v1.1
* Evaluable IMDC risk score
* Archival tumor specimen, and pretreatment tumor tissue from fresh biopsy at screening, if clinically feasible. Both archival and fresh samples are preferred.
* KPS score of >=70
* Recovery to baseline or Grade </= 1 NCI CTCAE v5.0 from toxicities related to any prior treatments, unless adverse events are clinically nonsignificant and/or stable in the opinion of the investigator. Grade 2 alopecia is allowed for study participation
* Adequate hematologic and end-organ function
* Negative HIV test at screening
* Negative hepatitis B testing at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Treatment with anti-cancer therapy within 14 days prior to initiation of study treatment
* Patients received cabozantinib at any time prior to screening
* Patients who received more than one ICI treatment in the locally advanced or metastatic setting
* Patients who received more than two prior lines of therapy in the locally advanced or metastatic setting
* Patients who have received a mammalian target of rapamycin (mTOR) inhibitor in any setting
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* History of malignancy other than renal carcinoma within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Radiotherapy for RCC within 14 days prior to Day 1 of Cycle 1
* Active tuberculosis
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after final dose of atezolizumab and 4 months after final dose of cabozantinib
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion of the investigator, could impact patient safety
* Pharmacologically uncompensated, symptomatic hypothyroidism
* Uncontrolled hypertension defined as sustained blood pressure >150 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment (all countries except France); sustained BP > 140 mmHg systolic or > 90 mmHg diastolic despite optimal antihypertensive treatment (France only)
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, unstable arrhythmia, or unstable angina) within 3 months prior to initiation of study treatment
* Significant vascular disease (e.g., aortic aneurysm or arterial dissection requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of Cycle 1
* History of congenital QT syndrome
* History or presence of an abnormal ECG that is clinically significant in the investigator's opinion
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitor dabigatran, direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g. clopidogrel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2025-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (125):
- United States (23):
  - University of Arizona, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Health System, La Jolla, California
  - UCLA, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Center - Denver, Littleton, Colorado
  - Woodlands Medical Specialists, P.A., Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - Memorial Sloan Kettering - Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - New York Oncology Hematology,P.C.-Albany, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology - Central South, Austin, Texas
  - University Of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists - Gainsville, Gainesville, Virginia
- Argentina (4):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Inst. Alexander Fleming, Buenos Aires
  - Hospital Britanico, Ciudad Autonoma Bs As
  - Centro Medico Austral OMI, Ciudad Autonoma Buenos Aires
- Australia (3):
  - Orange Hospital, Orange, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Bendigo Cancer Centre, Bendigo, Victoria
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- Herlev Hospital, Herlev, Denmark
- France (7):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Hopital Europeen Georges Pompidou, Paris
  - ICANS, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Zeisigwaldkliniken Bethanien, Chemnitz
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Krankenhaus Martha-Maria Halle-Dölau, Klinik für Urologie, Halle
  - Uniklinik-Eppendorf, Hamburg
  - Med. Hochschule Hannover, Hämatologie, Hämostaseologie, Onkologie u. Stammzelltransplantation, Hanover
  - Klinikum rechts der Isar der TU München, München
  - Universitaetsklinikum Muenster, Münster
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Greece (5):
  - Alexandras General Hospital of Athens, Athens
  - Attikon University General Hospital, Athens
  - Athens Medical Center, Athens
  - University Hospital of Larissa, Larissa
  - Diavalkaniko Hospital, Thessaloniki
- Italy (13):
  - A.O. Universitaria Ospedale Consorziale Policlinico Di Bari, Bari, Apulia
  - Istituto Tumori Napoli, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Policlinico Universitario "Agostino Gemelli", Rome, Lazio
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Fondazione Salvatore Maugeri, Pavia, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Fondazione del Piemonte per l?Oncologia (IRCCS), Candiolo (TO), Piedmont
  - Ospedale Di Macerata, Macerata, The Marches
  - Azienda Ospedaliera S. Maria - Terni, Terni, Umbria
  - A.O.U di Verona Policlinico G.B. Rossi, Verona, Veneto
- Japan (8):
  - Hokkaido University Hospital, Hokkaido
  - University of Tsukuba Hospital, Ibaraki
  - Yokohama City University Hospital, Kanagawa
  - Okayama University Hospital, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Tokushima University Hospital, Tokushima
  - Keio University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
- Poland (8):
  - Centrum Terapii Wspolczesnej J.M.Jasnorzewska Spolka Komandytowo-Akcyjna, ?ód?
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - SP ZOZ Wojewódzki Szpital Specjalistyczny nr 4, Bytom
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Szpital Kliniczny im. Heliodora ?wi?cickiego UM w Poznaniu, Późna
  - Szpital Grochowski im. dr med. Rafa?a Masztaka Sp. z o.o., Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - Dolno?l?skie Centrum Onkologii, Pulmonologii i Hematologii, Wroc?aw
- Russia (8):
  - St-Petersburg Regional Oncology Dispensary, Kuzmolovo, Leningrad
  - Branch of the company "Hadassah Medical LTD", Innovatsionnogo Tsentra Skolkovo, Moscow Oblast
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow, Moscow Oblast
  - SBIH "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of DHM", Moskva, Moscow Oblast
  - Private Healthcare Institution Clinical Hospital RZhD Medicine, Saint Petersburg, Sankt-Peterburg
  - AV Medical Ltd., Saint Petersburg, Sankt-Peterburg
  - Regional Clinical Oncology Hospital, Yaroslavl, Yaroslavl Oblast
  - Medical Center Avicenna, Novosibirsk
- South Korea (9):
  - Chungnam National University Hospital, Daejeon
  - CHA Bundang Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (20):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Hospital de Navarra, Navarra, Navarre
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Univ. Central de Asturias, Oviedo, Principality of Asturias
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro De Alcantara, Cáceres
  - Hospital Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Universitario la Fe, Valencia
- United Kingdom (4):
  - Royal Blackburn Hospital, Blackburn
  - Barts & London School of Med, London
  - Royal Marsden Hospital, London
  - Christie Hospital Nhs Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Pal SK, Albiges L, Tomczak P, Suarez C, Voss MH, de Velasco G, Chahoud J, Mochalova A, Procopio G, Mahammedi H, Zengerling F, Kim C, Osawa T, Angel M, Gupta S, Khan O, Bergthold G, Liu B, Kalaitzidou M, Huseni M, Scheffold C, Powles T, Choueiri TK. Atezolizumab plus cabozantinib versus cabozantinib monotherapy for patients with renal cell carcinoma after progression with previous immune checkpoint inhibitor treatment (CONTACT-03): a multicentre, randomised, open-label, phase 3 trial. Lancet. 2023 Jul 15;402(10397):185-195. doi: 10.1016/S0140-6736(23)00922-4. Epub 2023 Jun 5. PMID 37290461
- [Derived] Yang Y, Psutka SP, Parikh AB, Li M, Collier K, Miah A, Mori SV, Hinkley M, Tykodi SS, Hall E, Thompson JA, Yin M. Combining immune checkpoint inhibition plus tyrosine kinase inhibition as first and subsequent treatments for metastatic renal cell carcinoma. Cancer Med. 2022 Aug;11(16):3106-3114. doi: 10.1002/cam4.4679. Epub 2022 Mar 18. PMID 35304832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 147 locations in 15 countries: Argentina, Australia, Canada, Denmark, France, Germany, Greece, Italy, Japan, Republic of Korea, Poland, Russian Federation, Spain, United Kingdom, United States of America.
Groups:
- Cabozantinib (Control); Atezolizumab + Cabozantinib: Participants who received treatment until disease progression per RECIST v1.1, unacceptable toxicity, or symptomatic deterioration attributed to disease progression as determined by the investigator.
Period: Overall Study
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Started | 259 | 263
Received at Least One Dose of Study Treatment | 256 | 262
Completed (Early Discontinuation) | 157 | 161
Not Completed | 102 | 102
Not completed — Death | 86 | 89
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib | Total
Number analyzed (Participants) | 259 | 263 | 522
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 144 | 153 | 297
  >=65 years | 115 | 110 | 225
Age, Customized [Mean (Standard Deviation); unit: Number] | 61.8 (10.2) | 61.8 (9.9) | 61.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 59 | 121
  Male | 197 | 204 | 401
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 23 | 52
  Not Hispanic or Latino | 212 | 232 | 444
  Unknown or Not Reported | 18 | 8 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 23 | 33 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 2 | 8
  White | 213 | 219 | 432
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 16 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by an Independent Review Facility (IRF) (IRF-PFS) According to RECIST v1.1
Description: Progression Free Survival (PFS) is defined as the time from randomization to disease progression, as determined by the Independent Review Facility (IRF) per RECIST v1.1, or death from any cause, whichever occurs first. Data for patients who have not experienced disease progression or death were censored at the last tumor assessment date. Data for patients with no postbaseline tumor assessments were censored at the randomization date.
Time Frame: From randomization to the first occurrence of disease progression according to RECIST v1.1 (up to 2 years 5 months).
Population: The efficacy evaluable population included all patients who received at least one dose of each drug for their assigned treatment regimen.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 259 | 263
Months | 10.81 [9.95 to 12.45] | 10.55 [9.76 to 12.25]
Statistical Analysis 1: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Stratified Cox Proportional Hazards Model; p = 0.7844, Log Rank; Stratified; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.83 to 1.28] — Hazard ratios were estimated by Cox regression. If at least one stratum has <10 events at the time of analysis, the stratification factor that contains the level with the smallest number of patients will be removed from the stratified analysis
Statistical Analysis 2: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Cox Proportional Hazards Model; Test type: Other; p = 0.7195, Log Rank; Unstratified; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.84 to 1.29] — Hazard ratios were estimated by Cox regression

2. Primary Outcome: Overall Survival (OS)
Description: From randomization to death due to any cause. Data for patients who are not reported as having died at the date of analysis were censored at the date when they were last known to be alive. Patients who do not have post-baseline information were censored at the date of randomization.
Time Frame: From randomization to death due to any cause (up to 2 years 5 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 259 | 263
Months | NA [21.13 to NA] — Not estimable due to too few events having occurred. | 25.72 [21.52 to NA] — The upper limit of the 95% CI was not estimable because too few events had occurred.
Statistical Analysis 1: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Stratified Cox Proportional Hazards Model; p = 0.6902, Log Rank; Stratified; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.70 to 1.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Cox Proportional Hazards Model; p = 0.7853, Log Rank; Unstratified; Hazard Ratio (HR) = 0.96, 95% CI [0.71 to 1.27] — Hazard ratios were estimated by Cox regression

3. Secondary Outcome: Progression Free Survival (PFS) as Assessed by Investigators (INV-PFS), According to RECIST v1.1
Description: Progression Free Survival (PFS) is defined as the time from randomization to disease progression, as determined by the Investigators per RECIST v1.1, or death from any cause, whichever occurs first. Data for patients who have not experienced disease progression or death were censored at the last tumor assessment date. Data for patients with no postbaseline tumor assessments were censored at the randomization date.
Time Frame: From randomization to the first occurrence of disease progression according to RECIST v1.1 or death from any cause (whichever occurs first) (up to 2 years 5 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 259 | 263
Months | 10.41 [8.51 to 12.29] | 10.38 [8.41 to 10.94]
Statistical Analysis 1: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Stratified Cox Proportional Hazards Model; p = 0.8037, Log Rank; Stratified; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.83 to 1.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Cox Proportional Hazards Model; p = 0.7894, Log Rank; Unstratified; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.83 to 1.27] — Hazard ratios were estimated by Cox regression

4. Secondary Outcome: Investigator-assessed Overall Response Rate (ORR) (INV-ORR) According to RECIST v1.1
Description: Overall Response Rate (ORR) is defined as the proportion of participants who had an objective response (complete response [CR] or partial response [PR]) on two consecutive occasions at least 4 weeks apart according to RECIST v1.1. in the ORR evaluable population, defined as patients with measurable disease at baseline.
Time Frame: as for outcome 3
Population: The ORR evaluable population is defined as participants with measurable disease at baseline. There were discrepancies between the IRF and INV assessments of participants' measurable diseases at baseline, which are reflected in the number of participants analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 259 | 263
Percentage of Participants
  Responders (CR + PR) | 41.7 [35.63 to 47.96] | 38.0 [32.13 to 44.19]
  Complete Response (CR) | 0.8 [0.09 to 2.76] | 1.5 [0.42 to 3.85]
  Partial Response (PR) | 40.9 [34.88 to 47.18] | 36.5 [30.67 to 42.64]
  Stable Disease (SD) | 46.3 [40.14 to 52.61] | 48.3 [42.11 to 54.51]
  Progressive Disease (PD) | 6.6 [3.87 to 10.30] | 9.1 [5.93 to 13.27]
  Not Evaluable | 0 [0 to 1.4] | 0.8 [0.1 to 2.7]
  Missing | 5.4 [3 to 8.9] | 3.8 [1.8 to 6.9]
Statistical Analysis 1: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Difference in Overall Response Rates; p = 0.4306, Cochran-Mantel-Haenszel; Odds Ratio (OR) = -3.68, 95% CI 2-sided [-12.45 to 5.10] — Odds ratio 95% CI was constructed using the Wald method. If at least one stratum has <10 events at the time of analysis, the stratification factor containing the level with the smallest number of patients will be removed from the stratified analysis

5. Secondary Outcome: Independent Review Facility (IRF)-Assessed Overall Response Rate (ORR) (IRF-ORR) According to RECIST v1.1
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 254 | 259
Percentage of Participants
  Responders (CR + PR) | 40.9 [34.84 to 47.27] | 40.5 [34.51 to 46.79]
  Complete Response (CR) | 0.8 [0.10 to 2.82] | 0 [0.00 to 1.41]
  Partial Response (PR) | 40.2 [34.08 to 46.47] | 40.5 [34.51 to 46.79]
  Stable Disease (SD) | 47.6 [41.36 to 53.97] | 50.6 [44.32 to 56.82]
  Progressive Disease (PD) | 5.1 [2.75 to 8.59] | 4.2 [2.14 to 7.47]
  Not Evaluable | 0.8 [0.1 to 2.8] | 0.8 [0.1 to 2.8]
  Missing | 5.5 [3 to 9.1] | 3.9 [1.9 to 7]
Statistical Analysis 1: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Difference in Overall Response Rates; p = 0.9893, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.70 to 1.43] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Investigator-assessed Duration of Response (DOR) (INV-DOR) According to RECIST v1.1
Description: Duration of Response (DOR) is defined as the time from the first occurrence of a confirmed objective response (complete response [CR] or partial response [PR]) to disease progression, or death, whichever occurs first. Data for participants who have not experienced disease progression or death will be censored at the last tumor assessment date. If no tumor assessments were performed after the date of the first occurrence of CR or PR, data for DOR will be censored at the date of the first occurrence of CR or PR.
Time Frame: From the date of first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to 2 years 5 months)
Population: The DOR evaluable population is defined as participants with measurable disease at baseline who experienced a a confirmed objective response (complete response [CR] or partial response [PR]).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 108 | 100
Months | 12.19 [9.72 to 14.52] | NA [10.38 to NA] — Not estimable due to too few events having occurred.
Statistical Analysis 1: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Difference between Duration of Response (DOR) rates; p = 0.0816, Log Rank; Stratified; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.47 to 1.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Difference between Duration of Response (DOR) rates; p = 0.1099, Log Rank; Unstratified; Hazard Ratio (HR) = 0.72, 95% CI [0.49 to 1.08] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Independent Review Facility (IRF)-Assessed Duration of Response (DOR) (IRF-DOR) According to RECIST v1.1
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
Number analyzed (Participants) | 104 | 105
Months | 14.75 [11.30 to 20.01] | 12.65 [10.51 to 17.38]
Statistical Analysis 1: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Difference between Duration of Response (DOR) rates; p = 0.8354, Log Rank; Stratified; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.70 to 1.54] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cabozantinib (Control) vs Atezolizumab + Cabozantinib; Test type: Other — Difference between Duration of Response (DOR) rates; p = 0.8159, Log Rank; Unstratified; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.71 to 1.55] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All Adverse Event (AE) and Serious Adverse Event (SAE) data presented here were collected from date of randomization to primary completion date (up to 2 years 5 months). AE and SAE data continues to be collected until the end of the study and the results will be updated within 1 year of the final collection date.
Description: The incidence, nature, and severity of Adverse Events (AE) and Serious Adverse Events (SAE) were reported, with severity determined according to NCI CTCAE v5.0 of the safety population, defined as all randomized participants who received ≥1 dose of study treatment. All-Cause Mortality data are reported for the all-enrolled population. One participant enrolled but died before receiving study treatment.
Arm/Group | Cabozantinib (Control) | Atezolizumab + Cabozantinib
All-Cause Mortality (participants affected / at risk) | 87/259 | 89/263
Serious Adverse Events (participants affected / at risk) | 84/256 | 126/262
Other Adverse Events (participants affected / at risk) | 251/256 | 255/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (Control) (N=256) | Atezolizumab + Cabozantinib (N=262)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 3 (4)
Death (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 2 (2) | 1 (2)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 7 (7)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (2)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (3) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Aspergilloma (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (2) | 1 (1)
Febrile infection (Infections and infestations) | 1 (2) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Human herpesvirus 6 encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 4 (5)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5)
Vascular device infection (Infections and infestations) | 2 (3) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 4 (6)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 2 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (Control) (N=256) | Atezolizumab + Cabozantinib (N=262)
Anaemia (Blood and lymphatic system disorders) | 47 (64) | 52 (64)
Neutropenia (Blood and lymphatic system disorders) | 18 (35) | 15 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (33) | 21 (28)
Hypothyroidism (Endocrine disorders) | 97 (111) | 95 (115)
Abdominal pain (Gastrointestinal disorders) | 33 (41) | 14 (16)
Abdominal pain upper (Gastrointestinal disorders) | 17 (17) | 25 (27)
Constipation (Gastrointestinal disorders) | 42 (46) | 37 (44)
Diarrhoea (Gastrointestinal disorders) | 179 (340) | 170 (313)
Dyspepsia (Gastrointestinal disorders) | 20 (24) | 26 (31)
Nausea (Gastrointestinal disorders) | 92 (131) | 76 (98)
Stomatitis (Gastrointestinal disorders) | 43 (48) | 50 (66)
Vomiting (Gastrointestinal disorders) | 42 (77) | 36 (48)
Asthenia (General disorders) | 75 (88) | 75 (108)
Fatigue (General disorders) | 61 (83) | 71 (92)
Mucosal inflammation (General disorders) | 51 (70) | 45 (56)
Oedema peripheral (General disorders) | 12 (12) | 16 (16)
Pyrexia (General disorders) | 15 (20) | 32 (36)
COVID-19 (Infections and infestations) | 31 (32) | 36 (39)
Urinary tract infection (Infections and infestations) | 15 (19) | 23 (43)
Alanine aminotransferase increased (Investigations) | 57 (87) | 62 (93)
Aspartate aminotransferase increased (Investigations) | 61 (92) | 60 (87)
Blood alkaline phosphatase increased (Investigations) | 14 (15) | 17 (20)
Blood bilirubin increased (Investigations) | 13 (24) | 11 (14)
Blood creatinine increased (Investigations) | 16 (23) | 22 (24)
Blood lactate dehydrogenase increased (Investigations) | 11 (13) | 15 (19)
Blood thyroid stimulating hormone increased (Investigations) | 14 (14) | 17 (17)
Weight decreased (Investigations) | 64 (78) | 46 (51)
Decreased appetite (Metabolism and nutrition disorders) | 97 (119) | 99 (122)
Hyperkalaemia (Metabolism and nutrition disorders) | 15 (24) | 4 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (18) | 19 (22)
Hypocalcaemia (Metabolism and nutrition disorders) | 18 (27) | 19 (27)
Hypokalaemia (Metabolism and nutrition disorders) | 29 (39) | 26 (40)
Hypomagnesaemia (Metabolism and nutrition disorders) | 46 (62) | 37 (61)
Hypophosphataemia (Metabolism and nutrition disorders) | 26 (35) | 22 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (31) | 29 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 23 (24)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 14 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 18 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (24) | 14 (15)
Dizziness (Nervous system disorders) | 9 (10) | 23 (28)
Dysgeusia (Nervous system disorders) | 38 (43) | 39 (40)
Headache (Nervous system disorders) | 27 (31) | 27 (34)
Insomnia (Psychiatric disorders) | 13 (13) | 19 (20)
Proteinuria (Renal and urinary disorders) | 41 (52) | 40 (57)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 29 (35)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 37 (42)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 21 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (25) | 10 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 18 (22)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 8 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (23) | 11 (13)
Hair colour changes (Skin and subcutaneous tissue disorders) | 19 (19) | 9 (9)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 105 (130) | 101 (133)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (21) | 21 (23)
Rash (Skin and subcutaneous tissue disorders) | 27 (32) | 33 (41)
Hypertension (Vascular disorders) | 86 (103) | 70 (78)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Collaborators are Exelixis and Chugai. The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04338269/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04338269/SAP_001.pdf